CLINICAL TRIAL: NCT00558909
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 4 Weeks Treatment With Three Selected Oral Doses of BI 44847 as Tablet in Female and Male Patients With Type 2 Diabetes.
Brief Title: 4 Weeks Treatment of Type II Diabetic Patients With BI 44847
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1224.4
Record Dates: First submitted 2007-08-30; First posted 2007-11-15 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: BI 44847
Drug: placebo for BI 44847

SUMMARY:
The primary objective of the current study is to investigate the safety and tolerability of BI 44847 in male and female patients with type 2 diabetes following oral administration of repeated doses of 100 mg b.i.d, 400 mg b.i.d. and 800 mg b.i.d. over 28 days.

A secondary objective is the exploration of the pharmacokinetics and pharmacodynamics of BI 44847 after multiple dosing, including assessment of steady state.

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal or hysterectomised female patients with proven diagnosis of type 2 diabetes mellitus treated with diet and exercise only or with one or 2 oral hypoglycaemic agent other than glitazones. In case of 2 oral hypoglycaemic agents, at least one of these may be taken at no more than 50% of its maximum dose;
* Age = > 21 and Age = <70 years (female hysterectomised and male patients);
* Age = >55 and Age = <70 years (female postmenopausal patients);
* BMI = >18.5 and BMI = <40 kg/m2 (Body Mass Index);
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation.

Exclusion Criteria:

* Treatment with insulin, glitazones, or more than one oral hypoglycaemic agent (except if 2 agents and at least one of them not taken at more than 50% of maximum dose);
* Fasted blood glucose > 240 mg/dl on two consecutive days during wash-out; HbA1c > 8.5 % at screening;
* Clinically relevant concomitant diseases other than type 2 diabetes, hyperlipidaemia and medically treated hypertension;
* History of relevant allergy/hypersensitivity;
* Marked baseline prolongation of QT/QTc interval;
* History of additional risk factors for TdP;
* Any laboratory value outside the reference range and the clinical relevance is not acceptable in the opinion of the investigator, or the value is more than 3 times higher than the upper limit of the reference range;
* Concomitant medication except for acetylsalicylic acid, statins, antihypertensives (diuretics not allowed), beta-blockers for BPH and occasional use of paracetamol (doses of no more than 1000 mg; no more than 2000 mg per day; no more than 2 days per week);
* Change of drug dosing of allowed co-medication < the last 6 weeks; Intake of any medication < 5 half-lives of the respective drug prior to first administration of study medication or during the trial, except allowed co-medication;
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval (based on the knowledge at the time of patient inclusion) < 10 days prior to first administration of study medication or during the trial;
* Use of grapefruit (or its juice) < 10 days prior to first administration of study medication or during the trial;
* Participation in another trial with an investigational drug < two months prior to first administration of study medication or during the trial; Smoker;
* Inability to refrain from smoking on specified trial days; Alcohol abuse;
* Drug abuse;
* Blood donation;
* Excessive physical activity;
* Male patients not using adequate contraception;
* Women of childbearing potential, positive pregnancy test or lactating

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Weight and waist circumference - change from baseline | Day 28 (Hour = 647:30)
Frequency of patients with maximal increase from baseline QTcF and QTcB interval | 4 weeks
Frequency of patients with possible clinically significant abnormalities | 4 weeks
Micturition total frequency - change from baseline | Day 28
Global tolerability - number of patients by category | 4 weeks

SECONDARY OUTCOMES:
Cmax (maximum concentration of the analyte in plasma) | Day 1
Tmax (time from dosing to maximum concentration) | Day 1
t1/2 (terminal half-life of the analyte in plasma) | Day 1
λz (terminal rate constant in plasma) | Day 1
C12,1 (concentration of analyte in plasma at 12 hours post-drug administration after administration of the first dose) | Day 1
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point within the first dosing interval) | Day 1
AUC0-12 (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 12 h after administration of the first dose) | Day 1
Ae0-12 (amount of analyte that is eliminated in urine over the time interval 0 h to 12 h) | Day 1
fe0-12 (fraction of analyte excreted unchanged in urine from time points 0 h to 12 h) | Day 1
CLR (renal clearance of the analyte in plasma after extravascular administration - based on 0 - 12 hour data) | Day 1
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | Day 1
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Day 1
Cmax,ss (maximum concentration of the analyte in plasma at steady state over a uniform dosing interval) | Day 28
Cmin,ss (minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval) | Day 28
Cpre,N (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N) | Day 28
Cpre,ss (predose concentration of the analyte in plasma at steady state immediately before administration of the last dose) | Day 28
C12,ss (concentration of analyte in plasma at 12 hours post-drug administration at steady state) | Day 28
tmax,ss (time from dosing to maximum concentration at steady state) | Day 28
tmin,ss (time from dosing to minimum concentration during a dosing interval) | Day 28
AUC0-tz,ss (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point within the last dosing interval) | Day 28
AUC0-12,ss (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 12 h at steady-state) | Day 28
MRTpo,ss (mean residence time of the analyte in the body after 56 administrations (b.i.d.) at steady state) | Day 28
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | Day 28
Vz/F,ss (apparent volume of distribution during the terminal phase λz following an extravascular dose at steady state) | Day 28
Ae0-12,ss (amount of analyte that is eliminated in urine at steady state over the time interval 0 to 12 h) | Day 28
fe0-12,ss (fraction of analyte excreted unchanged in urine at steady state over the time interval 0 to 12 h) | Day 28
CLR,ss (renal clearance of the analyte at steady state - based on 0 - 12 hour data) | Day 28
RA,Cmax based on Cmax | following 55 doses (bid)
RA,AUC based on AUCτ | following 55 doses (bid)
Predose concentrations of the analyte in plasma | 5 minutes before drug administration on days 2,3,4,7,14,21,26,27,28 and 29
Change from baseline in UGE, AE0-24 | Day 27
Change from baseline in weighted MDG, AUEC0-24 | Day 27
Epre-corrected AUEC0-5 following OGTT | Day 28
Cavg (average concentration) | day 28
PTF (peak trough fluctuation). | day 28

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Germany (3):
  - 1224.4.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1224.4.49003 Boehringer Ingelheim Investigational Site, Mainz
  - 1224.4.49001 Boehringer Ingelheim Investigational Site, Neuss
- 1224.4.31001 Boehringer Ingelheim Investigational Site, Zuidlaren, Netherlands